CLINICAL TRIAL: NCT03904238
Title: Psychosocial Adjunctive Treatment for Hypersomnia (PATH): A Pilot Trial
Brief Title: Psychosocial Adjunctive Treatment for Hypersomnia (PATH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jason Ong, Associate Professor, Northwestern University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00207253; 185-SR-17 (Other Grant/Funding Number: American Academy of Sleep Medicine Foundation)
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Narcolepsy; Idiopathic Hypersomnia
Keywords: Hypersomnia; narcolepsy; idiopathic hypersomnia; psychosocial; cognitive-behavior therapy
MeSH Terms: conditions — Narcolepsy; Idiopathic Hypersomnia; Disorders of Excessive Somnolence | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants are assigned to receive CBT-H in one of two formats: 1) individually or 2) small groups. However, the contents of the intervention are the same.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-H (Individual format) (Experimental): Individual CBT-H consists of 6 weekly sessions that are conducted one-on-one with a study therapist using live videoconferencing or in-person. Each session is expected to last about 45 to 60 minutes.
  Interventions: Behavioral: Cognitive-Behavior Therapy for Hypersomnia (CBT-H)
- CBT-H (Group format) (Experimental): Group-based CBT-H consists of 6 weekly sessions that are conducted in groups with a study therapist using live videoconferencing or in-person. Each session is expected to last about 45 to 60 minutes. The treatment package consists of the same cognitive and behavioral modules as the individual CBT-H. However, participants are also provided the opportunity to share their experiences and provide peer support in the group format.
  Interventions: Behavioral: Cognitive-Behavior Therapy for Hypersomnia (CBT-H)

INTERVENTIONS:
Behavioral: Cognitive-Behavior Therapy for Hypersomnia (CBT-H) — The CBT-H intervention consists of 6 weekly sessions that are conducted either individually or in small groups. Each session is expected to last about 45 to 60 minutes and will be delivered a study therapist using live videoconferencing or in-person. The treatment package consists of cognitive and behavioral modules that include education about hypersomnia, coping skills training, emotion regulation regarding the perceived limitations of living with chronic hypersomnia (e.g., "I cannot live a full life because of my illness"), and behavioral techniques using scheduled naps, sleep hygiene, and regularizing sleep schedules at night which are on the current optional recommendations for hypersomnia.

SUMMARY:
Current pharmacological treatments for chronic hypersomnia (narcolepsy, idiopathic hypersomnia) can effectively reduce excessive daytime sleepiness but a high proportion of patients experience depressive symptoms and poor health-related quality of life. Unfortunately, there are currently no psychosocial interventions that directly addresses this issue. Therefore, the overall goal of this project is to gather initial outcome data and work out methodological issues to determine if a future pragmatic clinical trial is warranted.

DETAILED DESCRIPTION:
Chronic hypersomnia (CH) is a serious and debilitating condition involving persistent excessive daytime sleepiness (EDS) and includes narcolepsy and idiopathic hypersomnia (IH). Currently, pharmacotherapy is the only empirically-validated treatment for reducing EDS in this patient population but the burden of long-term management and adverse effects of the medication lead to poor health-related quality of life (HRQoL) and elevations in depressive symptoms

Evidence-based psychosocial interventions have been developed in other areas to improve HRQoL related to chronic illnesses, such as cancer and chronic pain. These interventions typically involve a package of cognitive and behavioral techniques teaching coping skills (e.g., emotion-focused and problem-focused coping), behavioral management of the chronic illness symptoms (e.g., relaxation for pain management), and other strategies to improve psychosocial functioning (e.g., mindfulness). However, no such interventions have been developed or used for people with CH. Therefore, a major research gap exists for an empirically-validated psychosocial intervention which is aimed directly at improving emotional functioning and HRQoL for people with CH.

The purpose of this project is to develop a cognitive-behavioral treatment for hypersomnia (CBT-H) and conducting a feasibility trial of CBT-H. The specific aims for this project are to: 1) develop and refine a treatment protocol for CBT-H; 2) identify the optimal delivery format of CBT-H; and 3) gather feasibility data on recruitment, retention, and selection criteria for a future clinical trial. The overall significance of this project is to improve the quality of care for people with CH by using a psychosocial intervention with medical management of hypersomnia.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females age 18 and older.
2. Meets criteria for Narcolepsy (Type I or II) or Idiopathic Hypersomnia (IH).
3. Moderate to severe symptoms of depression.
4. Established standard care for CH at a sleep clinic.

Exclusion Criteria:

1. Hypersomnia not of central origin.
2. Current suicidal ideation or intent.
3. Uncontrolled medical conditions or physical limitations that require immediate medical treatment that would prevent ability to engage in the treatment protocol.
4. Inability to engage in the treatment protocol due to a psychiatric or cognitive issue.
5. Untreated moderate-to-severe sleep-related breathing disorder.
6. Unable to attend intervention sessions due to accessibility or availability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ) | Change from Baseline PHQ at 6 weeks (Post-treatment)
  The PHQ is a 9-item self-report scale of depressive symptoms that has been validated to assess the severity of depression in clinical practice. PHQ-9 cut scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe depression, respectively.

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS) Self Efficacy Scale | Baseline to post-treatment (6 weeks)
  Measures general self-efficacy, self-efficacy for managing emotions, self-efficacy for managing social interactions, self-efficacy for managing symptoms using Computer Adaptive Testing (CAT) with higher scores reflecting better self-efficacy.
Patient Reported Outcomes Measurement Information System (PROMIS) Depression Scale | Baseline to post-treatment (6 weeks)
  Measures depressive symptoms using Computer Adaptive Testing (CAT) with higher scores reflecting more anxiety symptoms.
Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety Scale | Baseline to post-treatment (6 weeks)
  Measures anxiety symptoms using Computer Adaptive Testing (CAT) with higher scores reflecting more anxiety symptoms.
Patient Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Scale | Baseline to post-treatment (6 weeks)
  Measures sleep disturbances using Computer Adaptive Testing (CAT) with higher scores reflecting more sleep disturbance.
Patient Reported Outcomes Measurement Information System (PROMIS) Sleep-Related Impairment Scale | Baseline to post-treatment (6 weeks)
  Measures sleep-related impairment using Computer Adaptive Testing (CAT) with higher scores reflecting worse outcomes.
Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue Scale | Baseline to post-treatment (6 weeks)
  Measures fatigue using Computer Adaptive Testing (CAT) with higher scores reflecting worse outcomes.
Patient Reported Outcomes Measurement Information System (PROMIS) Phyiscal Function Scale | Baseline to post-treatment (6 weeks)
  Measures physical function using Computer Adaptive Testing (CAT) with higher scores reflecting better physical function.
Epworth Sleepiness Scale (ESS) | Baseline to post-treatment (6 weeks)
  The ESS consists of eight questions rated from 0 to 3, with higher scores indicating greater likelihood of falling asleep. Total scores of 10 or greater reflect excessive daytime sleepiness.
Functional Outcomes of Sleep Questionaire (FOSQ) | Baseline to post-treatment (6 weeks)
  The FOSQ assesses the impact of sleepiness on daily behaviors and quality of life. It is comprised of 30 items divided into five subscales: activity level, vigilance, intimate and sexual relationships, general productivity, and social outcome. Items are rated from 1 to 4, with higher score reflecting better functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Circadian and Sleep Medicine, Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ong JC, Dawson SC, Mundt JM, Moore C. Developing a cognitive behavioral therapy for hypersomnia using telehealth: a feasibility study. J Clin Sleep Med. 2020 Dec 15;16(12):2047-2062. doi: 10.5664/jcsm.8750. PMID 32804069